CLINICAL TRIAL: NCT00797043
Title: A Clinical Outcomes Protocol of Photon/Proton Beam Radiation Therapy for Carcinoma of the Skin of the Head and Neck With Perineural Invasion
Brief Title: Photon/Proton Radiation Therapy for Carcinoma of the Skin of the Head and Neck
Acronym: SK01
Status: Terminated | Type: Observational
Why Stopped: Slow enrollment, feasibility issues
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: UFPTI 0606-SK01
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Malignant Neoplasm of Skin Head and Neck
Keywords: Carcinoma of the skin of the head and neck; Proton radiation; Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Photon/Proton Radiation Therapy: Data consolidation and analysis

SUMMARY:
The purpose of this study is to collect information from the questionnaire and your medical records to see what effects the proton radiation has on you and your cancer and collect and analyze morbidity outcomes: Incidence of xerostomia (dry mouth) and tumor control.

DETAILED DESCRIPTION:
Data collection will be obtained from the patient's medical records including initial evaluation, pathology report, dosimetry information, radiotherapy completion records and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Carcinoma of the skin of the head and neck region with incidental or symptomatic perineural invasion.
* Biopsy-proven squamous cell carcinoma.
* Will receive treatment with proton radiation.

Exclusion Criteria:

* Evidence of distant metastasis.
* Previous irradiation for head and neck cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at radiation oncology clinic
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2008-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Collect and analyze morbidity outcomes: Incidence of grade 3 or higher xerostomia (dry mouth) | 1 year following the completion of radiation therapy

SECONDARY OUTCOMES:
Collect and analyze tumor control outcomes. | When each patient has been followed for a minimum of 6 months and then again at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Roi Dagan, MD, MS, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] BALLANTYNE AJ, MCCARTEN AB, IBANEZ ML. THE EXTENSION OF CANCER OF THE HEAD AND NECK THROUGH PERIPHERAL NERVES. Am J Surg. 1963 Oct;106:651-67. doi: 10.1016/0002-9610(63)90074-6. No abstract available. PMID 14070757
- [Background] Cottel WI. Perineural invasion by squamous-cell carcinoma. J Dermatol Surg Oncol. 1982 Jul;8(7):589-600. doi: 10.1111/j.1524-4725.1982.tb00317.x. PMID 6749931
- [Background] Mendenhall WM, Parsons JT, Mendenhall NP, Brant TA, Stringer SP, Cassisi NJ, Million RR. Carcinoma of the skin of the head and neck with perineural invasion. Head Neck. 1989 Jul-Aug;11(4):301-8. doi: 10.1002/hed.2880110404. PMID 2753698
- [Background] Mendenhall WM, Parsons JT, Mendenhall NP, Million RR. T2-T4 carcinoma of the skin of the head and neck treated with radical irradiation. Int J Radiat Oncol Biol Phys. 1987 Jul;13(7):975-81. doi: 10.1016/0360-3016(87)90034-4. PMID 3597161
- [Background] Al-Othman MO, Mendenhall WM, Amdur RJ. Radiotherapy alone for clinical T4 skin carcinoma of the head and neck with surgery reserved for salvage. Am J Otolaryngol. 2001 Nov-Dec;22(6):387-90. doi: 10.1053/ajot.2001.28083. PMID 11713722
- [Background] Mendenhall WM, Amdur RJ, Williams LS, Mancuso AA, Stringer SP, Price Mendenhall N. Carcinoma of the skin of the head and neck with perineural invasion. Head Neck. 2002 Jan;24(1):78-83. doi: 10.1002/hed.10025. PMID 11774406
- [Background] Parsons JT, Bova FJ, Fitzgerald CR, Mendenhall WM, Million RR. Radiation optic neuropathy after megavoltage external-beam irradiation: analysis of time-dose factors. Int J Radiat Oncol Biol Phys. 1994 Nov 15;30(4):755-63. doi: 10.1016/0360-3016(94)90346-8. PMID 7960976
- [Background] Bhandare N, Monroe AT, Morris CG, Bhatti MT, Mendenhall WM. Does altered fractionation influence the risk of radiation-induced optic neuropathy? Int J Radiat Oncol Biol Phys. 2005 Jul 15;62(4):1070-7. doi: 10.1016/j.ijrobp.2004.12.009. PMID 15990010
- [Background] Mendenhall WM, Amdur RJ, Siemann DW, Parsons JT. Altered fractionation in definitive irradiation of squamous cell carcinoma of the head and neck. Curr Opin Oncol. 2000 May;12(3):207-14. doi: 10.1097/00001622-200005000-00005. PMID 10841192